CLINICAL TRIAL: NCT02123927
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Ascending Single Dose Study of the Safety, Tolerability and Pharmacokinetics of TAK-438 in Healthy Male Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of TAK-438 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438/CPH-001; U1111-1153-7002 (Other: World Health Organization)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Ascending Single Dose Study
Keywords: Drug therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (13):
- Step 1: TAK-438 1 mg (Experimental): TAK-438 1 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-438
- Step 2: TAK-438 5 mg (Experimental): TAK-438 5 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-438
- Step 3: TAK-438 10 mg (Experimental): TAK-438 10 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-438
- Step 4: TAK-438 20 mg (Experimental): TAK-438 20 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-438
- Step 5: TAK-438 40 mg (Experimental): TAK-438 40 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-438
- Step 6: TAK-438 80 mg (Experimental): TAK-438 80 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-438
- Step 7: TAK-438 120 mg (Experimental): TAK-438 120 mg, tablets, orally, once on Day 1.
  Interventions: Drug: TAK-438
- Steps 1-7: Placebo (Placebo Comparator): TAK-438 placebo-matching tablets, orally, once on Day 1.
  Interventions: Drug: Placebo
- Step 8A: TAK-438 10 mg (Experimental): TAK-438 10 mg, tablets, orally, under fasted conditions, once on Day 1, Period 1, followed by a 13 day washout period, followed by TAK-438 10 mg, tablets, orally, under fed conditions, once on Day 1, Period 2.
  Interventions: Drug: TAK-438
- Step 8 B: TAK-438 10 mg (Experimental): TAK-438 10 mg, tablets, orally, under fed conditions, once on Day 1, Period 1, followed by a 13 day washout period, followed by TAK-438 10 mg, tablets, orally, under fasted conditions, once on Day 1, Period 2.
  Interventions: Drug: TAK-438
- Step 9A: TAK-438 40 mg (Experimental): TAK-438 40 mg, tablets, orally, under fasted conditions, once on Day 1, Period 1, followed by a 13 day washout period, followed by TAK-438 40 mg, tablets, orally, under fed conditions, once on Day 1, Period 2.
  Interventions: Drug: TAK-438
- Step 9B: TAK-438 40 mg (Experimental): TAK-438 40 mg, tablets, orally, under fed conditions, once on Day 1, Period 1, followed by a 13 day washout period, followed by TAK-438 40 mg, tablets, orally, under fasted conditions, once on Day 1, Period 2.
  Interventions: Drug: TAK-438
- Steps 8 (A & B) and 9 (A & B): Placebo (Placebo Comparator): TAK-438 placebo-matching tablets, orally, once on Day 1, Period 1, followed by a 13 day washout period, followed by TAK-438 placebo-matching tablets, orally, once on Day 1, Period 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-438 — TAK-438 tablets
  Arms: Step 1: TAK-438 1 mg; Step 2: TAK-438 5 mg; Step 3: TAK-438 10 mg; Step 4: TAK-438 20 mg; Step 5: TAK-438 40 mg; Step 6: TAK-438 80 mg; Step 7: TAK-438 120 mg; Step 8 B: TAK-438 10 mg; Step 8A: TAK-438 10 mg; Step 9A: TAK-438 40 mg; Step 9B: TAK-438 40 mg
Drug: Placebo — TAK-438 placebo-matching tablets
  Arms: Steps 1-7: Placebo; Steps 8 (A & B) and 9 (A & B): Placebo

SUMMARY:
The primary purpose of this study was to evaluate the single dose safety and pharmacokinetics of TAK-438 in healthy Japanese men.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-438. TAK-438 is being tested to find a safe and well-tolerated dose and to assess how TAK-438 moves throughout the body. This study will look at lab results and side effects in people who took TAK-438. This study consisted of 2 sequential studies: a single rising dose study (Steps 1 to 7) and a food-effect study (Steps 8 and 9).

The study population for Steps 1 to 7 consisted of 12 participants; with 9 participants randomized to receive a single dose of TAK-438, and 3 participants to receive placebo. Participants in Steps 1 to 7 received a single dose of study drug after a 10-hour fast. The starting dose was 1 mg followed by administrations of 5, 10, 20, 40, 80, and 120 mg. Steps 8 and 9 consisted of 12 participants in a 2-sequence, 2-period crossover design. Four participants were to receive a single dose of TAK-438 and 2 participants were to receive a single dose of placebo on Day 1, in the fasted state, and 4 participants were to receive a single dose of TAK-438 and 2 participants were to receive a single dose of placebo on Day 1 in the fed state, followed by a second single dose of TAK-438 or placebo in the alternative fed state after a 13 day minimum washout period. Participants in Steps 8 randomized to receive TAK-438 will receive 10 mg and participants in Step 9 will receive 40 mg.

This single-centre trial was conducted in Japan. The overall time to participate in this study was up to 32 days depending on the Step assignment. Participants made 3 to 5 visits to the clinic, including one or two 8-day periods of confinement to the clinic, also depending on Step assignment. All participants made a final visit 15 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy adult male volunteer.
2. Is between 20 and 45 years old when giving their informed consent.
3. Is able to understand the consents of the study and to follow them.
4. Provides their written informed consent prior to their participation in this study.
5. Weighs at least 50 kg and has a body mass index (BMI) of 18.5 to 25.0 kg/m^2 at screening.
6. Has negative results for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen/antibody, and serological tests for syphilis.
7. Participant whom the investigator or subinvestigator judged to be eligible on the basis of subjective symptoms, objective findings, vital signs, electrocardiogram (ECG) findings, and results of laboratory tests obtained until before the study drug administration.

Exclusion Criteria:

1. Has undergone upper gastrointestinal resectioning or vagotomy.
2. Has hypoacidity or anacidity: intragastric pH ≥ 5.5 at X-ray fluoroscopic confirmation of detained position of a pH probe inserted to measure baseline intragastric pH values.
3. Has a history of previous and current acid-related diseases including reflux esophagitis, gastric ulcer, duodenal ulcer, non-erosive gastroesophageal reflux disease, Barrett's esophagitis or Zollinger-Ellison syndrome.
4. Is undergoing H. pylori eradication within 6 months before the initiation of the study drug administration.
5. Has an inappropriate history of previous and current diseases for study participation including hepatic or renal disorders, and cardiovascular, hematological, endocrine, metabolic, pulmonary, gastrointestinal, neurological, urological, immunological, or psychological diseases.
6. Has a history of drug and food allergy.
7. Has a history of illegal drug abuse or alcoholism within 5 years before the initiation of the study drug administration.
8. Has peripheral vessels being difficult.
9. Has undergone whole blood drawing of at least 200 mL within 4 weeks or 400 mL within 12 weeks prior to initiation of the study drug administration.
10. Has undergone whole blood drawing of at least 800 mL in total within 52 weeks prior to initiation of the study drug administration.
11. Has undergone apheresis drawing [plasma (including platelet poor plasma or platelet rich plasma) and platelet component collection] within 2 weeks prior to initiation of the study drug administration.
12. Is taking any prescriptions or over the counter (OTC) drugs within 4 weeks prior to the study drug administration.
13. Has taken any vitamins, herbal medicines, and supplements including St. John's wort, Ginseng, kava kava, ginkgo biloba, melatonin within 4 weeks prior to initiation of the study drug administration.
14. Has had grapefruit (juice and pulp), or caffeine- or alcohol-containing foods or drinks within 72 hr prior to initiation of the study drug administration.
15. Has received other study drugs within 16 weeks prior to initiation of the study drug administration.
16. Participants whom the investigator or subinvestigator judged to be ineligible for study participation.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AE) | Day 1 to Day 15
  Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 14 days after the last dose of study drug, or if a serious adverse event, within 30 days after the last dose of study drug.
Number of Participants With Potentially Clinically Significant Vital Sign Findings | Day 1 to Day 15
  Participants with at least one potentially clinically significant post-baseline vital sign finding. Vital signs included blood pressure, pulse, respiratory rate, and body temperature (armpit), body weight, and body mass index (BMI).
Change from Baseline in Body Weight | Day 1 to Day 15
Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings | Day 1 to Day 15
Number of Participants With Potentially Clinically Significant Laboratory Evaluation Findings | Day 1 to Day 15
  Laboratory tests for hematology, biochemistry, coagulation and urinalysis were be performed.
AUC(0-48): Area Under the Plasma Concentration-Time Curve From Time 0 to hour 48 for TAK-438 and TAK-438 metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  AUC(0-48) is a measure of the area under the plasma concentration-time curve from time 0 to 48 hours, calculated using the linear trapezoidal rule.
AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-438 and TAK-438 metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  (AUC(0-tlqc) is a measure of total plasma exposure to the drug from time 0 to time of the last quantifiable concentration (AUC[0-tlqc]).
AUMC(0-tlqc): Area Under the First Moment Plasma Concentration-time Curve from Time 0 (t1) to Time of the Last Quantifiable Concentration (tlqc) for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  AUMC(0-tlqc) is a measure of the area under the first moment plasma concentration-time curve from time 0 to time of the last quantifiable concentration (tlqc), calculated using the linear trapezoidal rule.
MRT(0-tlqc): Mean Residence Time from Time 0 (t1) to Time of the Last Quantifiable Concentration (tlqc) for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  MRT(0-tlqc) is a measure of the mean residence time from time 0 to time of the last quantifiable concentration (tlqc) calculated as MRT(0-tlqc)=AUMC(0-tlqc)/AUC(0-tlqc).
Cmax: Maximum Observed Plasma Concentration TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  Time to reach the maximum plasma concentration (Tmax), equal to time (hours) to Cmax.
AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  AUC(0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Terminal Elimination Rate Constant (λz) for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  Terminal elimination rate constant (λz) is the rate at which drugs are eliminated from the body.
Terminal Elimination Half-life (T1/2) for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  Terminal Phase Elimination Half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Apparent Clearance (CL/F) Pharmacokinetic Parameter for TAK-438F | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC(0-24), expressed in L/hr.
AUMC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  AUMC(0-inf) is a measure of the area under the first moment plasma concentration-time curve from time 0 to infinity, calculated as AUMC(0-tlqc) + lqc x tlqc/λz + lqc/λz^2.
MRT: Mean Residence Time for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose (0 hours) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours postdose
  Mean residence time, calculated as MRT=AUMC(0-inf)/AUC(0-inf).
Cumulative Urinary Excretion Ratio for TAK-438F and TAK-438F metabolites M-I and M-II | Day 1 predose and 0-6, 6-12, 12-24, 24-36 and 36-48 hours postdose
  The cumulative urinary excretion ratio is defined as the percentage of the dose excreted in the urine.

SECONDARY OUTCOMES:
24-Hour Intragastric pH Profile | Baseline and Day 1
  To obtain intragastric pH a portable pH measuring device with a miniature glass electrode that was calibrated using standard pH 4 and pH 7 solutions was placed in the stomach transnasally and its positioned confirmed by X-ray guidance. pH data was recorded electronically 8:30 AM to 9:10 AM of the following day every 10 seconds.
Total Amount of Serum Gastrin | Baseline at prospective time of dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post prospective dose and Day 1 predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose
Total Amount of Serum Pepsinogen I | Baseline at prospective time of dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post prospective dose and Day 1 predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose
Total Amount of Serum Pepsinogen Ii | Baseline at prospective time of dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post prospective dose and Day 1 predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 and 48 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda